CLINICAL TRIAL: NCT02456597
Title: A Novel Concept for Continuous Peripheral Nerve Block - Popliteal Region
Brief Title: A Novel Concept for Continuous Peripheral Nerve Block - Sciatic Nerve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kai Henrik Wiborg Lange (Other)
Responsible Party: Sponsor-Investigator, Kai Henrik Wiborg Lange, Head Of Research, Hillerod Hospital, Denmark
Organization: Hillerod Hospital, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: H-15000927
Record Dates: First submitted 2015-04-01; First posted 2015-05-28 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Pain
Keywords: Peripheral Nerve Blocks
MeSH Terms: conditions — Pain | interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lidocainhydrochlorid (Active Comparator): Lidocaine 20mg/ml, 15 ml injected perineural at the sciatic nerve
  Interventions: Drug: lidocainhydrochlorid
- Isotonic saline (Placebo Comparator): 0.9% Saline Solution, 15ml injected perineural at the contralateral sciatic nerve
  Interventions: Drug: Isotonic Saline

INTERVENTIONS:
Drug: lidocainhydrochlorid — Lidocaine injected through the novel Catheter
  Other Names: Lidocaine, Xylocaine
  Arms: lidocainhydrochlorid
Drug: Isotonic Saline — Isotonic saline injected through the novel Catheter
  Other Names: Saline
  Arms: Isotonic saline

SUMMARY:
To investigate the function of a novel catheter for continuous peripheral nerve blocks in the popliteal nerve: Two key issues are investigated 1) Successful primary placement and function of the catheter for continuous peripheral nerve blocks confirmed by a decrease in motor function following injection of local analgesics through the catheter; 2) The rate of displacement after standardized movement of the limb where the catheter for continuous peripheral nerve blocks is inserted.

DETAILED DESCRIPTION:
Although peripheral nerve blocks are known to provide superior postoperative analgesia. Continuous peripheral nerve block (CPNB) are not used to the extent they deserve. This is predominantly due to variable success rates. Furthermore, the existing techniques for placing catheters for CPNBs are technically complicated and time consuming.4,5 Major problems include difficult insertion of the catheter tip past the needle, difficult visualization of catheter advancement, secondary displacement of the local anesthetic (LA) injection orifice(s) and limited possibility of repositioning the catheter once it has been left in situ. We have developed a new catheter for CPNBs to address and overcome these limitations.

Hence, the new catheter should primarily provide precise initial placement of the catheter, less risk of secondary displacement and a possibility to readjust the new catheter at any time point after initial placement. Furthermore, in-plane ultrasound (US) visualization during the entire procedure and during readjustment should be possible. The new catheter should also provide a simple and rapid technique with few components. Initial proof of concept studies in cadavers are promising with success rates close to 100 % both for initial placement and readjustment

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age at Visit X.
2. ASA classification ≤ II
3. Written informed consent obtained from volunteer and ability for volunteer to comply with the requirements of the study.

Exclusion Criteria:

1. BMI ≥ 30
2. Previous or ongoing surgery, pain or other disability of investigated region.
3. Prescriptive drugs other than anti-contraceptive.
4. Sensory or neurologic deficits in the investigated region
5. Allergy to LA
6. Pregnancy, breastfeeding, or unwilling to practice birth control during participation in the study.-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Muscle force (dynamometer) change from baseline | an average of three months
  Decreased muscle force measured with a dynamometer after intervention

SECONDARY OUTCOMES:
Surface EMG (sEMG) change from baseline | an average of three months
  Decreased EMG response (mV) after intervention
Displacement of catheter (mm) change from initial placement | an average of three months
  Displacement of catheter in millimeters assessed by ultrasound
Cutaneous Sensory Mapping (Decreased sensibility in the region innervated by Tibial and Popliteal nerves) change from baseline | an average of three months
  Decreased sensibility in the region innervated by Tibial and Popliteal nerves

CONTACTS AND LOCATIONS:
Overall Officials: Christian Rothe, Principal Investigator — Nordsjaellands Hospital